CLINICAL TRIAL: NCT00391989
Title: A Phase II Multicenter Study on the Treatment of Adult de Novo Philadelphia Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL) With the Protein Tyrosine Kinase Inhibitor BMS-354825. EudraCT Number 2005-005107-42.
Brief Title: Treatment of Adult Ph+ LAL With BMS-354825
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1205
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoblastic Leukemia, Acute
Keywords: Ph+ Acute Lymphoblastic Leukaemia; Dasatinib; targeted therapy; Patients with Ph positive and or BCR ABL positive ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
The primary objective of the trial is to estimate the activity of BMS-354825 (Dasatinib) in de novo adult Ph+ ALL patients in terms of hematological complete remission (HCR) rate.

DETAILED DESCRIPTION:
This open label phase II study of Dasatinib will enroll adult de novo Ph+ ALL patients. A minimum of 48 cases will be required to complete the study. Accrual is expected to be completed in 18 months. The study will be considered completed for patients in HCR after completion of a total of 12 weeks of treatment. After completion patients will go off study and will be treated according to the best treatment option for Ph+ ALL patients in 1st HCR. The enrollment in the post-remissional phase of the current GIMEMA LAL protocol will be suggested.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ph+ and/or BCR/ABL+ ALL
* Age ≥18 years old
* De novo ALL (within 14 days from diagnosis)
* No prior treatment with any anti-leukemic drugs with the exception of steroids for no more than 14 days (including the 7-day pretreatment already scheduled in the protocol)
* WHO performance status ≤2
* Absence of central nervous system (CNS) leukemia
* Normal serum level of potassium, total calcium corrected for serum albumin magnesium and phosphorus, or correctable with supplements
* ALT and AST ≤2.5 x ULN or ≤5.0 x ULN if considered due to leukemia
* Alkaline phosphatase ≤2.5 x ULN unless considered to leukemia
* Serum bilirubin ≤2 x ULN
* Serum creatinine ≤3 x ULN
* Serum amylase ≤1.5 x ULN and serum lipase ≤1.5 x ULN
* Normal cardiac function
* Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Impaired cardiac function, including any one of the following:
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BMS-354825 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection)
* Use of therapeutic warfarin
* Acute or chronic liver or renal disease considered unrelated to leukemia
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM¬CSF) ≤1 week prior to starting study drug
* Patients who are currently receiving treatment with any of the medications listed in "Appendix F" and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. The medications listed in "Appendix F" have the potential to prolong the QT interval.
* Patients who have received any anti-leukemic agents and treatments including steroids for more than 14 days including 7 days pretreatment that is part of the protocol
* Patients who have received any investigational drug in the last 2 weeks
* Patients who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of BMS-354825). Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Non compliant to oral medication patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Foà, MD, PhD, Principal Investigator — Università degli Studi di Roma "La Sapienza", Dipartimento di Biotecnologie Cellulari ed Ematolgia
Locations (36):
- Italy (36):
  - Ospedale San Donato USL 8, Arezzo, Arezzo
  - Università degli Studi di Bari, Bari, Bari
  - Ist.Ematologia e Oncologia Medica L.e A. Seragnoli, Bologna, Bologna
  - Azienda Spedali Civili, Brescia, Brescia
  - Osp. Reg. A. Di Summa, Brindisi, Brindisi
  - Servizio di Ematologia - CTMO - ASL 8 P.O. Binaghi, Cagliari, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania, Catania
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro, Catanzaro
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara, Ferrara
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova, Genova
  - Ospedale Niguarda " Ca Granda", Milan, Milano
  - Sez. di medicina Interna Oncologia ed Ematologia, Modena, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Div. TERE, Napoli, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli, Napoli
  - Ematologia Università Federico II, Napoli, Napoli
  - Ospedale S. Luigi Gonzaga, Orbassano, Orbassano
  - Dip. Oncologico "La Maddalena", Palermo, Palermo
  - Div. di Ematologia - A.O. "V. Cervello", Palermo, Palermo
  - Università degli Studi di Palermo - A.U. Policlinico, Palermo, Palermo
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia, Pavia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara, Pescara
  - Istituto di Ematologia- Ospedale San Carlo, Potenza, Potenza
  - Ospedale S.Maria delle Croci, Ravenna, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria, Reggio Calabria
  - Ospedale S. Camillo, Rome, Rome
  - Ospedale S.Eugenio, Rome, Rome
  - Università Cattolica del Sacro Cuore, Rome, Rome
  - Università degli Studi di Roma "La Sapienza", Rome, Rome
  - Università degli Studi di Tor Vergata, Rome, Rome
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari, Sassari
  - Policlinico Universitario, Udine, Udine
  - Policlinico G.B. Rossi, Verona, Verona
  - Ospedale Sant'Anna-17, Ronciglione, Viterbo
  - Nuovo Ospedale "Torrette", Ancona
  - Presidio Ospedaliero "C. e G.Mazzoni", Ascoli Piceno
  - Ospedale Casa Sollievo della sofferenza, San Giovanni Rotondo

REFERENCES:
- [Derived] Foa R, Vitale A, Vignetti M, Meloni G, Guarini A, De Propris MS, Elia L, Paoloni F, Fazi P, Cimino G, Nobile F, Ferrara F, Castagnola C, Sica S, Leoni P, Zuffa E, Fozza C, Luppi M, Candoni A, Iacobucci I, Soverini S, Mandelli F, Martinelli G, Baccarani M; GIMEMA Acute Leukemia Working Party. Dasatinib as first-line treatment for adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2011 Dec 15;118(25):6521-8. doi: 10.1182/blood-2011-05-351403. Epub 2011 Sep 19. PMID 21931113
- [Derived] Messina M, Chiaretti S, Iacobucci I, Tavolaro S, Lonetti A, Santangelo S, Elia L, Papayannidis C, Paoloni F, Vitale A, Guarini A, Martinelli G, Foa R. AICDA expression in BCR/ABL1-positive acute lymphoblastic leukaemia is associated with a peculiar gene expression profile. Br J Haematol. 2011 Mar;152(6):727-32. doi: 10.1111/j.1365-2141.2010.08449.x. Epub 2011 Jan 31. PMID 21623761

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: All patients registered in the study.
Period: Overall Study
Arm/Group | Study Group
Started | 55
Completed | 53
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib: All patients registered in the study.
Arm/Group | Dasatinib
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: Years] | 53.61 [23.79 to 76.49]
Gender [Count of Participants; unit: Participants]
  Female | 27
  Male | 26
White Blood Cells [Median (Full Range); unit: *10^9 cells/L] | 18.80 [2.20 to 132.90]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hematological Complete Remission (HCR) Obtained During the BMS Induction Treatment Within Day +85 From the Start of BMS (i.e., Whenever Achieved From the Start of the Experimental Drug).
Time Frame: End of the study, up to day 85
Measure: Number; unit: Patients
Arm/Group | Study Group
Number analyzed (Participants) | 53
Patients | 53

2. Secondary Outcome: The Incidence of Grade >2 CTC-NCI Side Effects and Toxicities;
Time Frame: End of study
Reporting Status: Not Posted

3. Secondary Outcome: The Best Cytogenetic Response Obtained During BMS Treatment Within Day +85, Whenever Achieved From the Start of the Experimental Drug;
Time Frame: End of study
Reporting Status: Not Posted

4. Secondary Outcome: the Best Molecular Response Obtained During BMS Treatment Within Day +85, Whenever Achieved From the Start of the Experimental Drug;
Time Frame: End of study
Reporting Status: Not Posted

5. Secondary Outcome: DFS, Defined as the Time Interval Between the Evaluation of HCR and Hematological Relapse of the Disease or Death in First HCR;
Time Frame: End of study
Reporting Status: Not Posted

6. Secondary Outcome: the Cumulative Incidence of Relapse;
Time Frame: End of study
Reporting Status: Not Posted

7. Secondary Outcome: OS, Defined as the Time Interval Between Inclusion and Death for Any Cause.
Time Frame: End of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 25 months.
Description: Physicians reporting whenever a SAE happened.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 13/53
Other Adverse Events (participants affected / at risk) | 12/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=53)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight gain (General disorders) | 1
Diarrhea (General disorders) | 1
Hypertransaminasemia (General disorders) | 1
Fever (General disorders) | 1
Proteinuria (General disorders) | 1
Increase of liver function (General disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Infection (Gastrointestinal disorders) | 1
Mood alteration (General disorders) | 1
hyperkalemia (General disorders) | 1
Nausea (General disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=53)
Fever (General disorders) | 1
Weight gain (General disorders) | 1
proteinuria (General disorders) | 1
Mild increase of liver function (General disorders) | 2
Gastrointestinal (Gastrointestinal disorders) | 1
Infection (General disorders) | 1
Mood alteration (General disorders) | 1
Hyperkalemia (General disorders) | 1
Acute pulmonary edema (General disorders) | 1
Diarrhea (General disorders) | 1
Hypertransaminasemia (General disorders) | 1
Nausea (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No